CLINICAL TRIAL: NCT01187654
Title: Comparison the Therapeutic Outcomes of Bone Marrow Derived AC 133+ and Mono-Nuclear Cells (MNC) Implantation in Patient With Acute Myocardial Infarction Underwent PCI Procedure
Brief Title: Bone Marrow Derived AC 133+ and Mono-Nuclear Cells (MNC) Implantation in Myocardial Infarction (MI) Patient
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Royan-Heart-002
Record Dates: First submitted 2010-08-18; First posted 2010-08-24 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2010-08

CONDITIONS: Myocardial Infarction
Keywords: myocardial infarction; bone marrow stem cell; AC133; mono nuclear cell
MeSH Terms: conditions — Myocardial Infarction | interventions — AC133 Antigen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AC133 recipients (Experimental): intra coronary injection of bone marrow derived AC133+ cells
  Interventions: Biological: AC133
- MNC recipients (Experimental): intra coronary injection of bone marrow derived MNC
  Interventions: Biological: MNC
- control (Active Comparator): injection of autologous serum
  Interventions: Biological: CONTROL

INTERVENTIONS:
Biological: AC133 — intra coronary injection of bone marrow derived AC133+ cells
  Other Names: AC133 injection
  Arms: AC133 recipients
Biological: MNC — intra coronary injection of bone marrow derived MNC
  Other Names: MNC injection
  Arms: MNC recipients
Biological: CONTROL — autologous serum injection
  Other Names: placebo injection
  Arms: control

SUMMARY:
Although a percutaneous coronary intervention (PCI) can be used to open up the blocked artery and restore blood flow to the heart muscle after myocardial infarction, there may be a significant amount of heart tissue that has been irreversibly damaged. Recent studies have shown that adult stem cells from bone marrow may be able to improve heart function and prevent from heart remodeling due to heart failure.

This study will evaluate the safety and effectiveness of using adult bone marrow derived stem cells for improving heart function in MI patients with Left Anterior Descending (LAD) involvement.

DETAILED DESCRIPTION:
Patient from both gender, who had acute MI within recent 3 Weeks in LAD territory and would underwent PCI are eligible for this study. The bone marrow derived AC 133+ and MNC would be intracoronary injected to the patients during PCI procedure. The control group would be received just serum during PCI. The patient would be followed every month and at the end of 6th and 18thmonth the case and control groups will be evaluated by stress echo and Tc99 scan.

The totality of evidence from trials investigating autologous whole bone marrow infusion into patients following myocardial infarction supports the safety of this approach in terms of efficacy

ELIGIBILITY:
Inclusion Criteria:

* BMI> 30
* First acute MI in LAD territory
* St elevation MI
* Ejection fraction: 20-45%
* at least two non - mobile or less mobile segment of left ventricular myocard.
* Successful PCI with stenting

Exclusion Criteria:

* Multivessel ceremony artery disease
* Pulmonary edema
* SBP < 80 mmHg
* Thrombocytopenia (PLT < 50, 000)
* INR > 2
* Hepatic failure or dysfunction
* Renal failure or dysfunction
* Positive HIV Ab/ HBC Ab/ HCV Ab/ HSV Ag
* Documental terminal illness
* Documental Malignancy
* Patient with sever coronary disease and unstability of vital sign
* History of leukopenia, Anemia, hepatic or renal dysfunction or malignancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-05; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Increase from baseline in ejection fraction | 6 months

SECONDARY OUTCOMES:
Decrease LVESV/LVEDV/LVM index | 6 months
  left ventricular end systolic volume (LVESV) left ventricular end diastolic volume (LVEDV) Left Ventricular mass (LVM)
Decrease the number of Non Viable segments from baseline | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Royan Institute; Masoud Ghassemi, MD, Principal Investigator — Royan Institute; Nasser Aghdami, PhD,MD, Study Director — Royan Institute; Davood Kazemi saleh, MD, Principal Investigator — Royan Institute; Hossein Baharvand, PhD, Principal Investigator — Royan Institute
Locations (1):
- Royan institute, Tehran, Iran